CLINICAL TRIAL: NCT03202498
Title: Safety and Tolerability of Yaq-001 in Patients With Cirrhosis ("CARBALIVE-SAFETY")
Brief Title: Safety and Tolerability of Yaq-001 in Patients With Cirrhosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic prevents patients from making in-hospital visits, which are mandatory to assessment of safety in this study
Sponsor: Yaqrit Ltd (Industry)
Collaborators: University College, London (Other); University of Brighton (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Azienda Ospedaliera di Padova (Other); Hospital Universitari Vall d'Hebron Research Institute (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); University of Lisbon (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); University of Bern (Other); Assistance Publique - Hôpitaux de Paris (Other); A2F Associates Limited (Other); Alpha Bioresearch S.L. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: Yaq001-S-001
Record Dates: First submitted 2017-04-05; First posted 2017-06-28 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-10

CONDITIONS: Liver Cirrhosis
Keywords: Cirrhosis, Liver; Fibrosis, Liver; Hepatic Cirrhosis; Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Cohort 1 (1:1 randomization):
  Standard medical treatment + Yaq-001 (4 g/ day) - n= 14.
  Standard medical treatment + placebo-control (placebo for 4 g of Yaq-001/ day) - n= 14.
  Cohort 2 (1:1 randomization):
  Standard medical treatment + Yaq-001 (8 g/ day) - n= 14.
  Standard medical treatment + placebo-control (placebo for 8 g of Yaq-001/ day) - n= 14.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (4g Yaq-001) (Experimental): Standard medical treatment + Yaq-001 (4 g/ day)
  Interventions: Device: 4g Yaq-001
- Cohort 1 (4g Placebo) (Placebo Comparator): Standard medical treatment + placebo-control (placebo for 4 g of Yaq-001/ day)
  Interventions: Other: 4g Placebo
- Cohort 2 (8g Yaq-001) (Experimental): Standard medical treatment + Yaq-001 (8 g/ day)
  Interventions: Device: 8g Yaq-001
- Cohort 2 (8g Placebo) (Placebo Comparator): Standard medical treatment + placebo-control (placebo for 8 g of Yaq-001/ day)
  Interventions: Other: 8g Placebo

INTERVENTIONS:
Device: 4g Yaq-001 — Study patients will be dosed daily with 4g of product Yaq-001 for a period of 12 weeks. The product will be provided as beads packed in individual sachets intended each for one oral administration. For each patient, the study duration will be up to 17 weeks, including the screening (up to 4 weeks), treatment (12 weeks) and 7-day follow up period.
  Arms: Cohort 1 (4g Yaq-001)
Other: 4g Placebo — Study patients will be dosed daily with a quantity of placebo equivalent to 4g of product Yaq-001 for a period of 12 weeks. The product will be provided as beads packed in individual sachets intended each for one oral administration. For each patient, the study duration will be up to 17 weeks, including the screening (up to 4 weeks), treatment (12 weeks) and 7-day follow up period.
  Arms: Cohort 1 (4g Placebo)
Device: 8g Yaq-001 — Study patients will be dosed daily with 8g of product Yaq-001 for a period of 12 weeks. The product will be provided as beads packed in individual sachets intended each for one oral administration. For each patient, the study duration will be up to 17 weeks, including the screening (up to 4 weeks), treatment (12 weeks) and 7-day follow up period.
  Arms: Cohort 2 (8g Yaq-001)
Other: 8g Placebo — Study patients will be dosed daily with a quantity of placebo equivalent to 8g of product Yaq-001 for a period of 12 weeks. The product will be provided as beads packed in individual sachets intended each for one oral administration. For each patient, the study duration will be up to 17 weeks, including the screening (up to 4 weeks), treatment (12 weeks) and 7-day follow up period.
  Arms: Cohort 2 (8g Placebo)

SUMMARY:
In patients with cirrhosis (scarring of the liver), bacterial fragments leak from the gut into the blood and cause harm. This study looks into a new way to lower the leakage of bacterial fragments into the blood.

Yaq-001 is a new type of carbon that in previous laboratory studies has been shown to have the ability to bind these bacterial fragments and so confine them to the gut. The purpose of this clinical trial is to test the product Yaq-001 for the first time in patients with cirrhosis.

This trial will assess if the treatment with Yaq-001 is safe, is well tolerated, and if it helps improve the overall health status of the cirrhotic patients.

Candidate patients must be at least 18 years old and have a clinical diagnosis of cirrhosis for any cause. Only postmenopausal women or with surgical sterilisation are eligible. Additional inclusion and exclusion criteria of medical nature will be determined with the investigator at the screening visit, by means of standard care routines plus an additional test to assess the bowel transit time.

Eligible patients will be randomly grouped to receive standard care treatment plus Yaq-001, or standard treatment plus placebo (non-active treatment). The use of placebo is necessary to better understand how safe and tolerable Yaq-001 really is.

The treatment lasts for 12 weeks. During treatment, the patient will be visited by a study doctor 5 times. At all the visits the patients will undergo a routine physical examination, electrocardiogram, collection of blood and urine samples. On three occasions the patients will be asked to provide additional samples of blood, urine and stool for analysis outside the hospital.

56 patients from 9 hospitals in UK, France, Italy, Portugal, Spain and Switzerland will participate in this study.

DETAILED DESCRIPTION:
First-in-human clinical investigation with Yaq-001. This is a multicentre, randomized, double blinded, placebo controlled trial to intended to evaluate safety and tolerability of oral administration of Yaq-001 therapy in two dosing cohorts.

56 cirrhotic patients with diuretic-responsive ascites will be enrolled. Patients will be randomized to two dosing cohorts.

Cohort 1 (1:1 randomization)

* Standard medical treatment + Yaq-001 (4 g/ day) - n= 14.
* Standard medical treatment + placebo-control (placebo for 4 g of Yaq-001/ day) - n= 14.

Cohort 2 (1:1 randomization)

* Standard medical treatment + Yaq-001 (8 g/ day) - n= 14.
* Standard medical treatment + placebo-control (placebo for 8 g of Yaq-001/ day) - n= 14.

Study patients will be dosed daily with Yaq-001 (or an equivalent quantity of placebo) for 12 weeks. Assessments of DSMB will take place after 4 and 12 weeks. Investigational centres specialized in the management of patients with liver cirrhosis will participate in the study.

For each patient, the study duration will be up to 17 weeks, including the screening (up to 4 weeks), treatment (12 weeks) and 7-day follow up period.

The total study duration is estimated to be approximately 6 months from screening of first patient until study completion of the last patient.

This project has received funding from the European Union's Horizon 2020 research and innovation programme under grant agreement No 634579.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients
2. Age ≥ 18 years at screening
3. Clinical diagnosis of cirrhosis for any cause. Liver biopsy is not required
4. Cirrhotic patients with diuretic-responsive ascites and Child-Pugh score = 7-11 inclusive
5. Abstinence from alcohol for at least 4 weeks prior to screening

Exclusion Criteria:

1. Refusal or inability (lack of capacity) to give informed consent
2. Prohibited medication within 4 weeks before the start of the study treatment: all oral antibiotics, immunosuppressants, long acting benzodiazepines or barbiturates and antiviral medication
3. Change in dose of proton pump inhibitor therapy within 4 weeks before the start of the study treatment
4. Patients with once daily medications in which orocaecal transit time is greater than 10 hours
5. Patients requiring medication in which the dosing schedule is three times per day or greater
6. Antiviral therapy for hepatitis C within 3 months prior to screening
7. Hospital admission for liver-related indication for at least 4 weeks (except paracentesis)
8. BMI > 35 or BMI < 18
9. Clostridium Difficile diarrhoea within 4 weeks before the start of the study treatment
10. Uncontrolled infection (chronic viral hepatitis is not an exclusion criterion)
11. Human immunodeficiency virus
12. Presence of a transjugular intrahepatic portosystemic shunt (TIPSS)
13. Participation in any clinical study of an investigational medicinal product within 30 days of five half-lives of the investigational product, whichever is longer
14. Presence of clinically relevant cardiovascular, pulmonary, gastro-intestinal, renal, hepatic, metabolic, haematological, neurological, psychiatric, systemic, ocular, gynaecologic or any acute infection disease or signs of acute illness that, in the opinion of the investigator, might compromise the patient's safe participation in the trial and/or results in a WHO performance status of 2 or more.
15. Presence of the history of cancer within the past 5 years with exception of hepatocellular carcinoma within Milan criteria, adequately treated localised basal cell carcinoma of the skin, in situ cervical carcinoma or solid malignancy surgical excised in total without recurrence for five years.
16. Women of child bearing potential. Only postmenopausal women or with surgical sterilization will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Assessment of reported and observed Serious Adverse Events | Day 1
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Day 1
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Day 1
  The percentage of patients who withdraw due to an AE will be tabulated by arm.
Assessment of reported and observed Serious Adverse Events | Week 1
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Week 1
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Week 1
  The percentage of patients who withdraw due to an AE will be tabulated by arm.
Assessment of reported and observed Serious Adverse Events | Week 4
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Week 4
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Week 4
  The percentage of patients who withdraw due to an AE will be tabulated by arm.
Assessment of reported and observed Serious Adverse Events | Week 8
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Week 8
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Week 8
  The percentage of patients who withdraw due to an AE will be tabulated by arm
Assessment of reported and observed Adverse Events | Week 12
  The percentage of patients experiencing SAEs will be tabulated by arm.
Assessment of treatment-related Serious Adverse Events | Week 12
  The percentage of patients experiencing device-related SAEs will be tabulated by arm.
Assessment of withdrawals due to Adverse Events | Week 12
  The percentage of patients who withdraw due to an AE will be tabulated by arm.

SECONDARY OUTCOMES:
Assessment of changes in blood endotoxin activity | The EAA will be performed at randomization, 1-week, 4-week, 8-week and 12-week visits.
  The changes from baseline in blood endotoxin activity, measured by the EAA, will be used as device-related performance indicator.
Assessment of changes in organ function as per the CHILD-PUGH score | CHILD-PUGH scores will be calculated at screening, randomization, 1-week, 4-week, 8-week and 12-week visits.
  Changes from baseline in kidney, liver, brain, intestinal and immune functions will be assessed by means of the CHILD-PUGH score.
Assessment of changes in organ function as per the MELD score | MELD scores will be calculated at screening, randomization, 1-week, 4-week, 8-week and 12-week visits.
  Changes from baseline in kidney, liver, brain, intestinal and immune functions will be assessed by means of the MELD score.
Assessment of changes in nutritional status | Global assessment will be performed at randomization, 1-week, 4-week, 8-week and 12-week visits.
  Changes from baseline in nutritional status be assessed by means of the global assessment score (RFH-GA);

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Jalan, Study Chair — Head, Liver Failure Group ILDH, Division of Medicine UCL Medical School Royal Free Campus Rowland Hill Street London NW32PF; Jane Macnaughtan, Study Director — Consultant, Liver Failure Group, ILDH, Division of Medicine UCL Medical School Royal Free Campus Rowland Hill Street London NW32PF
Locations (9):
- Hospital Beaujon, Hepatology and Liver Intensive Care,, Clichy, France
- Italy (2):
  - Policlinico S.Orsola Malpighi, Department of Medical and Surgical Sciences, Bologna
  - Azienda Ospedaliera di Padova, Hepatic Emergencies Unit, Padua
- University Hospital of Santa Maria, Lisbon, Portugal
- Spain (3):
  - Hospital Vall d'Hebron, Liver Unit, Barcelona
  - Hospital Clinic of Barcelona , Liver Unit,, Barcelona
  - Hospital Ramon y Cajal, Department of Gastroenterology and Hepatology, Madrid
- Inselspital Universitaet Bern, Department for Visceral Surgery and Medicine,, Bern, Switzerland
- Royal Free Hospital, Institute of Liver and Digestive Disease, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu J, MacNaughtan J, Kerbert AJC, Portlock T, Martinez Gonzalez J, Jin Y, Clasen F, Habtesion A, Ji H, Jin Q, Phillips A, De Chiara F, Ingavle G, Jimenez C, Zaccherini G, Husi K, Rodriguez Gandia MA, Cordero P, Soeda J, McConaghy L, Oben J, Church K, Li JV, Wu H, Jalan A, Gines P, Sola E, Eaton S, Morgan C, Kowalski M, Green D, Gander A, Edwards LA, Cox IJ, Cortez-Pinto H, Avery T, Wiest R, Durand F, Caraceni P, Elosua R, Vila J, Pavesi M, Arroyo V, Davies N, Mookerjee RP, Vargas V, Sandeman S, Mehta G, Shoaie S, Marchesi J, Albillos A, Andreola F, Jalan R. Clinical, experimental and pathophysiological effects of Yaq-001: a non-absorbable, gut-restricted adsorbent in models and patients with cirrhosis. Gut. 2024 Jun 6;73(7):1183-1198. doi: 10.1136/gutjnl-2023-330699. PMID 38621924